CLINICAL TRIAL: NCT05615389
Title: A Pilot Study of Medicinal Cannabis in Paediatric Patients Undergoing Palliative Care for Non-oncological Conditions
Brief Title: Pilot Study of MC in Paediatric Palliative Care
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: RCH HREC 88284
Record Dates: First submitted 2022-11-07; First posted 2022-11-14 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Palliative Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medicinal Cannabis C12T12 (Experimental): C12T12 Ruby Balanced Oil (Cannatrek Ltd, Australia). 12.5mg/ml CBD and 12.5mg/ml THC in sunflower oil.
  Interventions: Drug: Medicinal Cannabis - C12T12
- Medicinal Cannabis C20T5 (Experimental): C20T5 Ruby CBD Oil (Cannatrek Ltd, Australia). 20mg/ml CBD and 5mg/ml THC in sunflower oil.
  Interventions: Drug: Medicinal Cannabis - C20T5

INTERVENTIONS:
Drug: Medicinal Cannabis - C12T12 — Participants randomised to receive C12T12 Ruby Balanced Oil will commence with 0.008ml/kg/day (0.1 mg/kg/day THC) in two divided doses, and titrate up in four steps (increase by 0.008ml/kg/day every four days) over 16 days up to a maintenance dose of 0.04ml/kg/day (0.5mg/kg/day THC) in two divided doses, with a ceiling dose of 2ml/day (25mg/day THC) for participants weighing 50kg or more. The maintenance dose will then be continued from day 17 until day 42.
  Down-titration will occur for 16 days after the end of study visit, in the reverse of the up-titration period.
  Arms: Medicinal Cannabis C12T12
Drug: Medicinal Cannabis - C20T5 — Participants randomised to the C20T5 Ruby CBD Oil will receive a matched volume to the C12T12 arm during the up-titration, maintenance, and down-titration phases.
  Arms: Medicinal Cannabis C20T5

SUMMARY:
The goal of this pilot study is to explore the feasibility and acceptability of a medicinal cannabis clinical trial into easing the symptoms of children undergoing palliative care for non-oncological conditions. The trial will evaluate the study design including recruitment strategy, medication tolerability, duration and outcomes to determine acceptability and feasibility for participating families. The data collected will then be used to design a full-scale multi-centre trial.

Participants will be randomly allocated to receive one of two medicinal cannabis products. Neither the participants nor researchers will know the study drug allocation until the end of the trial.

DETAILED DESCRIPTION:
This is a single site, double-blind, randomized, pilot study of 10 participants investigating two medicinal cannabis (MC) products in children aged 6 months to 21 years who are undergoing palliative care for non-oncological conditions. Eligible participants will be randomized 1:1 to receive one of two medicinal cannabis products (C12T12 or C20T5).

The primary objective of this pilot study is to evaluate all elements of the study design (recruitment strategy, study duration, study procedures, study medication tolerance and outcome measures) to assess if they are acceptable and feasible for the conduct of a full-scale randomised trial of MC to reduce symptom burden in paediatric patients undergoing palliative care for non-oncological conditions.

The secondary objective of this study is to collect preliminary data on the safety of two different oral MC oil formulations in this population.

Each participants will be involved in the trial for up to 100 days:

* Screening period: Up to 14 days
* Up-titration: day 1 to day 16
* Maintenance treatment period: day 17 to day 42
* Down-titration: day 43 (end of maintenance period clinic visit) to day 58
* Post-treatment follow-up: day 59 to day 86.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 6 months to 21 years of age;
2. Receiving care in the Victorian Paediatric Palliative Care Program for a non-oncological condition;
3. Pain, dystonia and/or gut dysfunction parent-rated symptom score above threshold, defined by rating on the relevant revised Memorial Symptom Assessment Scale (MSAS) question(s) of:

   1. Frequency: "Frequently" or "Almost Constantly", AND
   2. Severity: "Moderate", "Severe", or "Very Severe", AND
   3. Distress: "Quite a bit", or "Very much";
4. No changes in medication or other interventions in the two weeks prior to randomization;
5. Participant and family have the ability to comply with the protocol requirements, in the opinion of the investigator;
6. Agrees not to drive for the duration of the study.

Exclusion Criteria:

1. Non-English speaking parents.
2. Participant history of psychosis, schizophrenia, bipolar disorder, or major depressive disorder, or a first degree family history of psychosis.
3. Taking medications which are known to interact with medicinal cannabis: warfarin, mTOR inhibitors (e.g sirolimus, tacrolimus), anti-cancer agents, citalopram >20mg/day, escitalopram >10mg/day.
4. Abnormal liver function tests defined as ALT > 3 x ULN
5. Current use of illicit drugs or medicinal cannabis, or use in the 4 weeks prior to screening
6. Pregnant or intending to become pregnant during the study, or breastfeeding.
7. History of clinically significant suicidal thoughts in the prior 12 months.
8. Life expectancy less than 3 months in the opinion of the investigators
9. Allergy to any of the components in the investigatory products (eg sunflower oil)
10. Diagnosis of a malignant condition

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Study participant recruitment completion time, calculated as the time required to reach a sample size of 10. | From the date of pre-screening the first participant until the tenth participant is randomized, up to 2 years.
  The time taken to complete recruitment will be calculated as the number of months from the date of commencing recruitment to the date of randomizing the tenth participant.
Participant withdrawal rate, calculated as the number of participants who withdraw from the trial as a proportion of the total number of participants randomized. | Day 1 to day 43 (date of the end of the maintenance dosing period clinic visit)
  The number of participants who withdraw from the trial will be calculated as a proportion of the total number of participants randomized.
Study medication tolerability, as indicated by the proportion of participants who tolerate the protocol dosing schedule. | Day 1 to day 43 (date of the end of the maintenance dosing period clinic visit)
  The number of participants who adhere to the protocol dosing schedule without medication related protocol deviations, treatment discontinuations or dose modifications will be calculated as a proportion of the total sample for each arm (C12T12 and C20T5).
Participant adherence to the study medication dosing schedule, calculated as the proportion of participants who demonstrate acceptable medication compliance. | Day 58 (date of end of treatment)
  Medication compliance will be assessed through pharmacy calculations from returned bottle volumes. Acceptable compliance will fall within the range of 80-120%. The number of participants with acceptable medication compliance will be reported as a proportion of the total sample randomized.
Study visit attendance, calculated as the proportion of visits completed across the study sample. | Screening to day 43 (date of the end of the maintenance dosing period clinic visit)
  The number of study visits attended by all participants will be calculated as a proportion of the total possible visits in accordance with the study protocol.
Blood test completion, calculated as the proportion of blood tests completed across the study sample. | Screening to day 43 (date of the end of the maintenance dosing period clinic visit)
  The number of study blood tests completed by all participants will be calculated as a proportion of the total possible blood tests in accordance with the study protocol.
Parent questionnaire completion, calculated as the proportion of parent-report questionnaires completed across the study sample. | Screening to day 86 (participant trial completion)
  The number of study questionnaires completed by all parents will be calculated as a proportion of the total possible questionnaires requiring completion in accordance with the study protocol.
Self-report questionnaire completion, calculated as the proportion of adolescent self-report questionnaires completed across the study sample. | Screening to day 86 (participant trial completion)
  The number of study self-report questionnaires completed by all participants will be calculated as a proportion of the total possible questionnaires requiring completion in accordance with the study protocol.
Study design acceptability will be evaluated through a parent-completed study specific evaluation questionnaire completed at the end of the study. | Day 86 (participant trial completion)
  Study design acceptability will be assessed using an evaluation questionnaire developed specifically for this study, which uses Likert scales to assess satisfaction with recruitment, medication tolerability, frequency of study visits, burden of completing questionnaires, and overall study quality. Parents will complete this questionnaire at the end of their study participation (day 86). Data will be reported for each item individually, as the proportion of parents who responded positively on the Likert scale, where higher scores indicate more favorable responses.

SECONDARY OUTCOMES:
The frequency of adverse events as reported on the modified version of the Liverpool Adverse Event Profile (LAEP) at day 43 will be summarized across the two medicinal cannabis treatment arms. | Day 43 (date of the end of the maintenance dosing period clinic visit)
  Completed by the parent or guardian, the LAEP was designed to capture known side-effects of anti-epileptic medication. The modified version includes additional items to ascertain other known side-effects of medicinal cannabis. This measure includes 34 items. Adverse Events (AEs) reported on the LAEP will be considered significant if a 2-point increase in severity is reported from baseline to end of the maintenance dosing period (day 43). The frequency of AEs meeting this criteria will be presented for the two medicinal cannabis treatment arms respectively.
The frequency of adverse events as reported throughout the study will be summarized across the two medicinal cannabis treatment arms. | Day 1 to day 86 (participant trial completion)
  All possible adverse events will be recorded, as reported at study visits, during safety check phone calls and in between scheduled appointments. All Serious Adverse Events will be published, as well as all non-serious adverse events deemed by the investigators to be at least possibly related to the study drug. The frequency of these adverse events will be presented for the two medicinal cannabis treatment arms respectively.

CONTACTS AND LOCATIONS:
Overall Officials: A/Prof Daryl Efron, Principal Investigator — Murdoch Childrens Research Institute
Locations (1):
- Royal Children's Hospital / Murdoch Children's Research Institute, Parkville, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data set collected for this analysis of the Pilot Study of MC in Paediatric Palliative Care will be available six months after publication of the primary outcome. The study protocol and analysis plan will also be available. The data must be obtained from the Murdoch Children's Research Institute. Prior to releasing any data the following are required: a data access agreement must be signed between relevant parties, the 'Pilot Study of MC in Paediatric Palliative Care' Study Management Group must see and approve the data analysis plan describing how the data will be analysed, there must be an agreement around appropriate acknowledgment and any additional costs involved must be covered. Should the Study Management Group be unavailable, this role is delegated to the Murdoch Children's Research Institute. Data will only be shared with a recognized research organisation which has approved the proposed analysis plan.
Supporting Information: Study Protocol, SAP
Time Frame: 6 months after publication of primary outcome
Access Criteria: 1) Data access agreement; 2) approval by Trial Steering Committee; 3) recognized research institutions.